CLINICAL TRIAL: NCT00386503
Title: A Randomized, Open-Label, Cross-Over Study, to Compare the Bioavailability of the Fixed Combination of Amodiaquine and Artesunate (COARSUCAM™) After Single Oral Administration Under Fed and Fasted Conditions in Healthy Subjects
Brief Title: Bioavailability of the Fixed Combination of Amodiaquine and Artesunate Under Fed & Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARAMF_L_01570
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination

INTERVENTIONS:
Drug: Artesunate + Amodiaquine

SUMMARY:
* Primary Objective: to evaluate the interaction with food after a single oral dose of a fixed combination of amodiaquine (AQ) and artesunate (AS) (COARSUCAM™) in healthy male subjects
* Secondary Objective: to assess the clinical and biological safety and tolerability of Coarsucam™

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian subjects
* Weight between 50 kg and 90 kg. 18 ≤ Body Mass Index ≤ 28 kg/m2.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2006-06; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics/Time course of the plasma concentrations of AS, AQ & their pharmacologically active metabolites dihydroartemisinin (DHA) & desethylamodiaquine (DSA), used to determine:Tmax, Cmax, t1/2, AUC(0-t) & AUC(0-Inf) for AS, DHA & AQ | During all the study conduct
Tmax, Cmax, Truncated AUC(0-10d) for DSA | during the study conduct

SECONDARY OUTCOMES:
Safety and tolerability/Adverse events, physical examinations, vital signs including heart rate and blood pressure, ECG and laboratory parameters. | From the signature of the informed consent up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Lameyre, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France